CLINICAL TRIAL: NCT07131657
Title: A Phase II, Single Arm, Open-label, Three-dose Group Study to Evaluate the Efficacy and Safety of Ropivacaine-betamethasone-clonidine (Ropiclobet) Injectable Solution for Regional Anesthesia and Post-operative Pain Control in Patients Undergoing Upper Extremity Surgery Below Shoulder
Brief Title: Ropiclobet for Regional Anesthesia and Post-Operative Pain Control in Upper Extremity Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHARMAFINA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF_002
Record Dates: First submitted 2025-07-31; First posted 2025-08-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Nerve Block; Upper Extremity Surgery
Keywords: ropivacaine; clonidine; betamethasone; supraclavicular brachial nerve block
MeSH Terms: interventions — Ropivacaine; Clonidine; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nerve block arm (Experimental): Volunteers will undergo supraclavicular brachial nerve block preoperatively using the combination drug Ropiclobet (Ropivacaine-Clonidine-Betamethasone)
  Interventions: Drug: Ropivacaine + Clonidine + Betamethasone

INTERVENTIONS:
Drug: Ropivacaine + Clonidine + Betamethasone — Ropivacaine HCl - Betamethasone Sodium Phosphate - Clonidine HCl 5.0/0.4*/0.015 mg/mL (The solution contains 0.53 mg of betamethasone sodium phosphate, equivalent to 0.4 mg of betamethasone)
  Group I: A total of 20 mL will be injected: 10 mL Ropiclobet (1 ampoule) + 10 mL of 0.9% isotonic saline
Drug: Ropivacaine + Clonidine + Betamethasone — Ropivacaine HCl - Betamethasone Sodium Phosphate - Clonidine HCl 5.0/0.4*/0.015 mg/mL (The solution contains 0.53 mg of betamethasone sodium phosphate, equivalent to 0.4 mg of betamethasone)
  Group II: A total of 20 mL will be injected: 15 mL Ropiclobet (1.5 ampoules) + 5 mL of 0.9% isotonic saline
Drug: Ropivacaine + Clonidine + Betamethasone — Ropivacaine HCl - Betamethasone Sodium Phosphate - Clonidine HCl 5.0/0.4*/0.015 mg/mL (The solution contains 0.53 mg of betamethasone sodium phosphate, equivalent to 0.4 mg of betamethasone)
  Group III: A total of 20 mL will be injected: 20 mL Ropiclobet (2 ampoules)

SUMMARY:
This is a national, single-center, single-arm, open-label Phase II clinical trial designed to evaluate the efficacy and safety of Ropiclobet, a fixed-dose injectable solution containing Ropivacaine HCl, Betamethasone Sodium Phosphate, and Clonidine HCl.

The study includes three non-randomized dose groups and will enroll a total of 60 adult volunteers undergoing upper extremity surgery (arm, elbow, forearm, or hand). All participants will receive a single administration of Ropiclobet via supraclavicular brachial plexus block (SCB) under ultrasound guidance. Sedation may be provided if necessary; however, participants requiring general anesthesia will be excluded from the study.

Postoperatively, volunteers will be monitored in the PACU for 2 hours, followed by transfer to a regular hospital ward under anesthesiology supervision. All participants will remain under clinical observation for 48 hours following the procedure. If the sensory or motor block persists beyond this period, monitoring will continue until full resolution and an additional 6 hours of observation will be provided. Follow-up visits are scheduled for Day 15 and Day 30 post-procedure.

The primary efficacy endpoint is the duration of analgesia and the primary safety endpoint is the incidence and characterization of all adverse events occurring during the procedure and within 30 days postoperatively.

DETAILED DESCRIPTION:
This national, single-center, single-arm, open-label Phase II clinical trial includes three dose groups and aims to evaluate the efficacy and safety of Ropiclobet. Ropiclobet Injectable Solution is a fixed-dose combination containing Ropivacaine HCl, Betamethasone Sodium Phosphate, and Clonidine HCl at concentrations of 5.0/0.4*/0.015 mg/mL (*the 10 mL ampoule contains 0.53 mg of betamethasone sodium phosphate, equivalent to 0.4 mg of betamethasone).

A total of 60 volunteers (Hospitalized patients in the orthopedic department or outpatients who are scheduled for surgery) undergoing upper extremity surgery (including arm, elbow, forearm, and hand surgeries) will receive a single administration of the Ropiclobet combination via supraclavicular brachial nerve blockade (SCB) under ultrasound guidance.

The study will include three dose groups:

* Group I: 10 mL Ropiclobet combination (1 ampoule) diluted with 10 mL of 0.9% isotonic saline
* Group II: 15 mL Ropiclobet combination (1.5 ampoules) diluted with 5 mL of 0.9% isotonic saline
* Group III: 20 mL Ropiclobet combination (2 ampoules), administered undiluted. There will be no randomization for dose groups. The first 20 participants will be assigned to Group I. The study team will assess safety and efficacy parameters in these participants. Following the completion of 20 participants in Group I, the study will proceed to Group II. Group III will follow in the same manner, with 20 participants planned per group.

Ropiclobet injection will be performed preoperatively under sterile conditions by an experienced anesthesiologist. Only sedation may be administered if needed, and volunteers requiring general anesthesia will be withdrawn from the study.

Standard monitoring will include ECG, non-invasive blood pressure measurement, and pulse oximetry. Postoperatively, volunteers will be monitored in the PACU for 2 hours, followed by observation in the hospital ward under an anesthesiologist's supervision. Volunteers will remain under clinical observation for 48 hours post-procedure. If motor or sensory blockade persists beyond this period, monitoring will continue until full resolution plus an additional 6 hours. Follow-up visits will be at Day 15 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age of ≥18 years and ≤ 65 years at the time of consent.
* Ability and willingness to provide informed consent or consent from their legal representative and willingness to comply with all planned visits and study procedures.
* American Society of Anesthesiologists (ASA) physical status class of I-III
* BMI ≤ 30 kg/m2
* An ECG within normal values or clinically insignificant findings.
* Patients undergoing upper extremity procedures suitable for SCB anesthesia, including arm, elbow, forearm, and hand surgeries.
* Emergency and/or elective surgeries
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy testing at screening visit.

Exclusion Criteria:

* An inability to cooperate during the block placement.
* Patients undergoing shoulder procedures.
* History of allergy to active ingredients (including their derivatives) of the study medication.
* History of allergy to analgesics (e.g. acetaminophen, non-steroidal anti-inflammatory medications, oral opioid analgesics)
* History of shoulder or clavicular surgery.
* Known bronchopulmonary or phrenic pathology compromising respiratory function.
* Existing chronic pain disorders or history of use of ≥ 30mg oxycodone or equivalent per day
* Pre-existing neurological deficits or peripheral neuropathy involving the operative upper extremity
* Infection at the puncture site for the block.
* History of coagulopathy disorders and/or bleeding diathesis.
* Pregnant or breastfeeding.
* History of any documented medical condition considered to be clinically significant and could potentially affect patient safety or study outcome, in the opinion of the investigator: uncontrolled diabetes, uncontrolled hypertension, cardiovascular diseases, acute or chronic kidney diseases, liver diseases, psychiatric disorders, malignancy, systemic infection.
* Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening which, in the opinion of the investigator, may put the patient at risk because of his/her participation in the study, or might influence the results of the study, or the patient's ability to complete the entire duration of the study.
* Participation in a clinical trial involving current or another investigational product in the previous 3 months.
* Currently taking long-term systemic steroids (excluding inhaled medication for asthma treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | From end of Ropiclobet injection to the first sensation of pain at surgical site (minutes/hours), up to 48 hours
Number of treatment-related adverse events assessed by NCI-CTCAE | From the beginning of the nerve block procedure to the end of study visit at 30 days

SECONDARY OUTCOMES:
Pain at rest | pre-block, and 0, 2, 4, 6, 12, 18, 24 and 48 hours post-block, on Day 15 and 30.
  Assessment of pain at rest using the Visual Analog Scale (VAS), 0-10 scale (0 (no pain) to 10 (worst possible pain))
Pain during movement | pre-block, and 0, 2, 4, 6, 12, 18, 24 and 48 hours post-block, on Day 15 and 30
  Assessment of pain during movement of the surgical site using Visual Analog Scale (VAS), 0-10 scale (0 (no pain) to 10 (worst possible pain))
Onset time of motor block | Pre-block, and at 5, 10, 15, 20, 25, 30 minutes, as well as 6, 12, 24 and 48 hours post-injection.
  Onset time of motor block is defined as the time (hour/minutes) from the completion of Ropiclobet injection to the onset of motor block. This will be assessed by grip strength test.
Duration of motor block | From nerve block procedure to the resolution of the motor block, up to 48 hours
  The time of resolution of the motor block (in minutes or hours), assessed by grip strength tests.
Onset time of sensory block | Pre-block, and at 5, 10, 15, 20, 25, 30 minutes, as well as 6, 12, 24 and 48 hours post-injection.
  Onset time of sensory block is defined as the time (hour/minutes) from end of Ropiclobet injection to the onset of sensory block. This will be assessed by cold and touch tests across C5-C8 dermatomes.
Duration of sensory block | From nerve block procedure to the resolution of the sensory block, up to 48 hours
  The time of resolution of the sensorial block (in minutes or hours)
Required rescue analgesia | Perioperative (from nerve block procedure to the end of surgery)
  Assessment of the frequency of required rescue analgesia intra-operatively.
Required rescue analgesia | From the end of surgery up to 48 hours
  Assessment of the frequency of required rescue analgesia postoperatively
Patient satisfaction | 24 hours following nerve block procedure, and on Day 15 and 30
  assessment of patient satisfaction using Visual Analog Scale (VAS), 0-10 scale (0=worst, 10=best)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No